CLINICAL TRIAL: NCT02089828
Title: Randomized Control Trial on Purified CD34+ Cells Versus Peripheral Blood Mononuclear Cells in Treatment of Critical Limb Ischemia
Brief Title: Purified CD34+ Cells Versus Peripheral Blood Mononuclear Cells in Treatment of Critical Limb Ischemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2014-021
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Thromboangiitis Obliterans; Arteritis; Peripheral Arterial Disease
MeSH Terms: conditions — Thromboangiitis Obliterans; Arteritis; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- autologous purified CD34+ cell (Experimental): transplantation of autologous purified CD34+ cell
  Interventions: Other: autologous purified CD34+ cells
- autologous PB-MNC (Active Comparator): transplantation of autologous peripheral blood mononuclear cells
  Interventions: Other: autologous peripheral blood mononuclear cells

INTERVENTIONS:
Other: autologous purified CD34+ cells
  Arms: autologous purified CD34+ cell
Other: autologous peripheral blood mononuclear cells
  Arms: autologous PB-MNC

SUMMARY:
To compare the efficacy and cost-effectiveness between purified CD34+ cells and peripheral blood mononuclear cells in treatment of critical limb ischemia

ELIGIBILITY:
Inclusion Criteria:

* Rutherford scale of 4-5
* thromboangiitis obliterans, peripheral arterial disease, or arteritis caused by other etiologies, such as collagen diseases
* surgical or endovascular procedures are considered unlikely to have successful long-term revascularization, or have failed
* more than 4 weeks of critical limb ischemia
* if present, a non-healing ulcer after more than 4 weeks of optimal care by a wound care physician and a nurse

Exclusion Criteria:

* within 3 months of an acute myocardial infarction
* any contraindication for the administration of granulocyte colony stimulating factor (G-CSF)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
major-amputation-free survival rate | at 6 months

SECONDARY OUTCOMES:
improvement on transcutaneous partial oxygen pressure | at 3 months

OTHER OUTCOMES:
improvement on peak pain-free walking time | at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Fu, M.D., Study Director — Fudan University; Zhihui Dong, M.D., Principal Investigator — Fudan University
Locations (1):
- Zhihui Dong, Shanghai, China

REFERENCES:
- [Background] Dong Z, Chen B, Fu W, Wang Y, Guo D, Wei Z, Xu X, Mendelsohn FO. Transplantation of purified CD34+ cells in the treatment of critical limb ischemia. J Vasc Surg. 2013 Aug;58(2):404-411.e3. doi: 10.1016/j.jvs.2013.01.037. Epub 2013 Apr 21. PMID 23611711
- [Derived] Liu H, Pan T, Liu Y, Fang Y, Fang G, Jiang X, Chen B, Wei Z, Gu S, Liu P, Fu W, Dong Z. The peripheral blood mononuclear cells versus purified CD34+ cells transplantation in patients with angiitis-induced critical limb ischemia trial: 5-year outcomes and return to work analysis-a randomized single-blinded non-inferiority trial. Stem Cell Res Ther. 2022 Mar 21;13(1):116. doi: 10.1186/s13287-022-02804-4. PMID 35313967
- [Derived] Liu H, Pan T, Fang Y, Fang G, Liu Y, Jiang X, Chen B, Wei Z, Gu S, Liu P, Fu W, Dong Z. Three-year outcomes of peripheral blood mononuclear cells vs purified CD34+ cells in the treatment of angiitis-induced no-option critical limb ischemia and a cost-effectiveness assessment: A randomized single-blinded noninferiority trial. Stem Cells Transl Med. 2021 May;10(5):647-659. doi: 10.1002/sctm.20-0033. Epub 2021 Jan 5. PMID 33399273
- [Derived] Dong Z, Pan T, Fang Y, Wei Z, Gu S, Fang G, Liu Y, Luo Y, Liu H, Zhang T, Hu M, Guo D, Xu X, Chen B, Jiang J, Yang J, Shi Z, Zhu T, Shi Y, Liu P, Fu W. Purified CD34+ cells versus peripheral blood mononuclear cells in the treatment of angiitis-induced no-option critical limb ischaemia: 12-Month results of a prospective randomised single-blinded non-inferiority trial. EBioMedicine. 2018 Sep;35:46-57. doi: 10.1016/j.ebiom.2018.08.038. Epub 2018 Aug 29. PMID 30172703